CLINICAL TRIAL: NCT04756934
Title: A Phase I Study of Tolerance and Pharmacokinetics of HX008 (a Humanized Monoclonal Antibody Targeting PD-1) Plus LP002 (a Humanized Monoclonal Antibody Targeting PD-L1) in Patients With Locally Advanced or Metastatic Melanoma Who Have Experienced Progressed Disease in Previous Anti-PD-1 or PD-L1 Therapy.
Brief Title: A Study of HX008 Plus LP002 for the Treatment of Patients With Advanced Melanoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taizhou HoudeAoke Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LP002-LH001
Record Dates: First submitted 2021-02-08; First posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Ia: LP002 dose escalation-1mg/kg (Experimental): 3-6 participants will receive HX008 of 200mg, Q3W plus LP002 of 1mg/kg, Q3W for up to 1 year.
  Interventions: Drug: HX008; Drug: LP002
- Ia: LP002 dose escalation-3mg/kg (Experimental): 3-6 participants will receive HX008 of 200mg, Q3W plus LP002 of 3mg/kg, Q3W for up to 1 year.
  Interventions: Drug: HX008; Drug: LP002
- Ia: LP002 dose escalation-5mg/kg (Experimental): 3-6 participants will receive HX008 of 200mg, Q3W plus LP002 of 5mg/kg, Q3W for up to 1 year.
  Interventions: Drug: HX008; Drug: LP002
- Ib: Expansion (Experimental): Approximately 30 participants will receive HX008 of 200mg, Q3W plus LP002 of the recommended dose, Q3W for up to 1 year.
  Interventions: Drug: HX008; Drug: LP002
- Ib: Control (Experimental): Approximately 15 participants will receive LP002 of recommended dose, Q3W for up to 1 year.
  Interventions: Drug: LP002

INTERVENTIONS:
Drug: HX008 — HX008: 200mg, Q3W
  Arms: Ia: LP002 dose escalation-1mg/kg; Ia: LP002 dose escalation-3mg/kg; Ia: LP002 dose escalation-5mg/kg; Ib: Expansion
Drug: LP002 — LP002: 1mg/kg, or 3mg/kg, or 5mg/kg, Q3W

SUMMARY:
The subsequent treatment choices for the patients with advanced melanoma, who have failed the immune checkpoint inhibitor therapy of single agent. Evidences showed that PD-1 and PD-L1 signalling pathways are not redundant. Blocking both of them could produce synergistic effect. HX008 and LP002 are humanized monoclonal antibodies targeting PD-1 on T cells and PD-L1 on tumor cells respectively. In this study, participants with locally advanced or metastatic melanoma who have failed previous anti-PD-1 or PD-L1 will be administrated with HX008 plus LP002. The safety and preliminary efficacy will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent voluntarily. Understand this protocol and be willing and able to adhere to the study visit schedule.
* Male and Female aged 18 to 75 are eligible.
* Histologic diagnosis of locally advanced or metastatic melanoma, who are unable to undergo complete resection, while ocular melanoma is excluded, and the overall rate of mucosal melanoma is no more than 22%.
* Has experienced progressed disease in previous anti-PD-1 or PD-L1 therapy for the locally advanced or metastatic melanoma (anti-PD-1 or PD-L1 therapy as neo-adjuvant or adjuvant therapy could be accepted if progressed disease occured with 6 months after the last dose of treatment).
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Life expectancy ≥ 3 months.
* With at least 1 measurable extracranial lesion based on RECIST v1.1, and no previous radiotherapy administrated to the measurable lesions.
* Central nervous system metastases must be asymptomatic with or without treatment, and be stable for at least 3 months based on CT/MRI, and no need for systemic steroids within 4 weeks prior to the first dose of the study drug.
* Provide with tumor specimen (for testing the expression of PD -L1).
* Has sufficient organ and bone marrow function to meet the following laboratory examination standards (without blood transfusion within 14 days prior to enrollment): neutrophils ≥ 1.5 x 10^9/L; white blood cells ≥3.0 x 10^9/L; platelets ≥ 100 x 10^9/L; hemoglobin ≥ 90 g/L; serum creatinine ≤1.5x ULN; aspartic transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN without, and ≤ 5 x ULN with hepatic metastasis; total bilirubin ≤ 1.5 x ULN; INR≤2 x ULN, aPTT≤1.5 x ULN (except for those undergoing anticoagulant therapy).
* Reproductive men and women of childbearing age are willing to take effective contraceptive measures from signing the informed consent form to 3 months after the last administration of the trial drug.

Exclusion Criteria:

* Prior malignancy active within the previous 5 years except for locally curable cancers that have been apparently cured, such as carcinoma in situ of the cervix or basal cell skin cancer.
* Has experienced severe immunotherapy related toxicity in the previous anti-PD-1 / PD-L1 monoclonal antibody treatment, including but not limited to: Grade 3 / 4 pneumonia, proteinuria, uveitis or upper scleritis, myasthenia gravis, pancreatitis, hepatitis, bullous skin diseases (including SJS, TEN); grade 2-4 encephalitis, myocarditis; any grade of Guillain Barre syndrome, transverse myelitis; severe inflammatory arthritis that significantly impact the quality of patient's life;
* Known to has BRAF V600 mutation before signing informed consent form, and has not received any corresponding targeted therapy.
* With adverse reactions of previous treatment that have not recovered to CTCAE V5.0 grade ≤ 1, except for the residual hair loss effect.
* With active or history of autoimmune diseases that may recur (e.g., systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease, multiple sclerosis, vasculitis, glomerulitis, etc.), or patients with high risk (e.g., organ transplantation requiring immunosuppressive therapy). While those with the following diseases were allowed to be enrolled: a) Stable patients with type I diabetes after a fixed dose of insulin; b) Autoimmune hypothyroidism requiring hormone replacement therapy only; c) Skin diseases requiring no systemic treatment (e.g. eczema, skin rash covering less than 10% of the body surface, psoriasis without ophthalmic symptoms, etc.).
* Expecting to receive major surgery during the study period including 4 weeks prior to the first dose of the study drug.
* Need to receive systemic corticosteroids (dose equivalent to > 10 mg prednisone / day) or other immunosuppressive drugs within 14 days before enrollment or during the study period. Those under the following conditions are eligible: a) Locally external use or inhaled corticosteroids; b) short-term (≤ 7 days) use of glucocorticoids for the prevention or treatment of non autoimmune allergic diseases.
* Has active digestive ulcer, incomplete intestinal obstruction, active gastrointestinal hemorrhage or perforation.
* Has active interstitial pneumonia, pulmonary fibrosis, acute pulmonary disorders, et al.
* Has uncontrolled systemic diseases, for instance, cardiovascular and cerebrovascular disease, diabetes, hypertension, tuberculosis.
* History of human immunodeficiency virus infection, acquired or congenital immunodeficiency disease, organ transplantation or stem cell transplantation.
* Has active chronic HBV or HCV infection, except those with HBV DNA viral load ≤500 IU/mL or <10^3 copies/mL, or HCV RNA negative after adequate treatment.
* Has severe infection within 4 weeks or active infection requiring IV infusion or oral administration of antibiotics within 2 weeks prior to the first dose of the study drug.
* Known to be allergic to macromolecular protein agents or monoclonal antibody; Known to has a history of severe allergies (CTCAE v5.0 ≥ grade 3) to any of the components in the study drug.
* Has participated in other clinical trial within 4 weeks prior to the first dose of the study drug.
* Alcohol dependence or drug abuse within recent one year.
* Has a history of confirmed neurological or mental disorders, such as epilepsy, dementia; or with poor compliance; or the presence of peripheral neurological disorders.
* Is pregnant or breastfeeding.
* Has received a live vaccine within 30 days prior to the first dose of trial treatment.
* Other reasons disqualifying the entering of this study based on the evaluation of the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2020-08-20 (Actual); Primary Completion 2021-08-20 (Estimated); Study Completion 2022-08-20 (Estimated)

PRIMARY OUTCOMES:
DLT (dose limited toxicity) rate | 6 months
  To observe how many participants experience DLT in each LP002 dose group in phase Ia.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 2 years
Objective Response Rate (ORR) | 1 year
  Percentage of subjects achieving complete response (CR) and partial response (PR).
Terminal half-life (T1 / 2) of HX008 and LP002 | 1 year
Area under curve (AUC) of HX008 and LP002 | 1 year
Apparent volume of distribution of HX008 and LP002 | 1 year
Systemic clearance of HX008 and LP002 | 1 year
Cmax of HX008 and LP002 | 1 year
Cmin of HX008 and LP002 | 1 year
Tmax of HX008 and LP002 | 1 year

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | 1 year
  Disease Control Rate (DCR) refers to the proportion of subjects who achieve CR, PR and SD through imaging evaluation.
Duration of Response (DOR) | 2 years
  Duration of Response (DOR) is defined as the time from the first evidence of response (PR or CR) to the first evidence of PD or the date of death for any reason.
Progression-Free Survival (PFS) | 2 years
  Progression-free survival (PFS) is defined as the time from the first study drug treatment to disease progression (PD) or to death of the subject due to any reason.
Overall survival (OS) | 2 years
  Overall survival (OS) refers to the time from the first study drug treatment to death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China